CLINICAL TRIAL: NCT00067847
Title: Evaluation of California's SB 19 Pupil Nutrition Act
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, Los Angeles (Other); University of California, Berkeley (Other); California Department of Education (Other); The California Endowment (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECSB19PNA (completed)
Record Dates: First submitted 2003-08-28; First posted 2003-09-01 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: obesity; food policy; physical fitness (Respiratory Burst); academic achievement
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: State-directed nutrition policy change

SUMMARY:
Four California school districts will be randomized to early implementation of California's SB 19 Pupil Nutrition Act or to business as usual. Over 5000 4th, 5th and 7th graders will be evaluated at baseline, 4-month, and 16-month follow-up in order to determine if the SB 19 nutrition and physical activity policies have had an impact on students' risk of excess body weight. The impact of early implementation of SB 19 on academic achievement will also be assessed.

DETAILED DESCRIPTION:
Four California school districts will be randomized to early implementation of California's SB 19 Pupil Nutrition Act or to business as usual.

The nutrition provisions in SB19 include assuring that NO elementary school sells carbonated beverages at any time and that no middle schools sell carbonated beverages until after the end of the lunch hour each day. The nutrition provisions also include some restrictions on the sale of high-fat, high-sugar snack foods as well as encouragement to make fruits and vegetables more available to students. The legislation further encourages school districts to invest more heavily in providing students with opportunities to be physically active. High schools are NOT affected by this legislation.

Over 5000 4th, 5th, and 7th graders from 28 schools will be evaluated at baseline, 4-month and 16-month follow-up in order to determine if the SB 19 nutrition and physical activity policies have had an impact on students' risk of excess body weight. The principal outcome measure is sex- and age-adjusted BMI percentile as determined from the CDC growthchart percentiles. Other measures include waist circumference, time to complete one mile run/walk, and blood pressure.

The impact of early implementation of SB 19 on academic achievement will also be assessed, using students' standardized math and language arts achievement test scores.

ELIGIBILITY:
healthy 4th, 5th or 7th graders able to fill out a 30-minute questionnaire in English and able to participate in aerobic physical activity.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5020
Dates: Start 2003-07; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: William J McCarthy, Ph.D., Principal Investigator — WestEd-Los Alamitos & UCLA Division of Cancer Prevention and Control Research
Locations (1):
- WestEd-Los Alamitos & UCLA Division of Cancer Prevention and Control Research, Los Angeles, California, United States

REFERENCES:
- See also: Dietary Guidelines for Americans (5th ed.) — http://www.health.gov/dietaryguidelines/
- See also: Legislative language of California's SB 19 Pupil Nutrition Act — http://www.leginfo.ca.gov/pub/01-02/bill/sen/sb_0001-0050/sb_19_bill_20011014_chaptered.pdf